CLINICAL TRIAL: NCT05193175
Title: Effects of Breaking up Sitting Time on Cardiometabolic Risk Markers and Cardiac Function Post Myocardial Infarction
Acronym: MOVE-MI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bedfordshire (Other)
Responsible Party: Principal Investigator, Abbie C. Bell, PhD Candidate, University of Bedfordshire
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 265468
Record Dates: First submitted 2021-12-06; First posted 2022-01-14 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Standing Position

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prolonged sitting (Experimental): Uninterrupted sitting for 6 hours.
  Interventions: Behavioral: Prolonged sitting
- Sitting interrupted with standing (Experimental): Sitting interrupted with 5 minutes of static standing every 30 minutes for 6 hours.
  Interventions: Behavioral: Prolonged sitting
- Sitting interrupted with light stepping (Experimental): Sitting interrupted with 5 minutes of light intensity stepping every 30 minutes using a metronome at the intensity determined during preliminary testing. This replicates active recovery time currently performed in a phase III CR class.
  Interventions: Behavioral: Prolonged sitting

INTERVENTIONS:
Behavioral: Prolonged sitting — Cross over design, where participants will take part in all three interventions listed above: 1) uninterrupted sitting, 2) sitting interrupted with standing and 3) sitting interrupted with light stepping
  Other Names: Sitting interrupted with standing; Sitting interrupted with light stepping

SUMMARY:
Cardiovascular Disease (CVD) is one of the greatest causes of mortality and morbidity globally, particularly in middle to high income countries. In the UK alone, it was accountable for 124,641 deaths in 2017. Further to this, CVD contributes to a vast economic burden, costing the National Health Service (NHS) £19billion annually. This is mainly due to a significant number of hospital readmissions following a first cardiac event (198,000 per annum).

Following a cardiac event, an individual is therefore recommended to reduce their risk factors, including lipid profile, smoking status and physical inactivity, to reduce their risk of a secondary event. In healthy individuals, regularly breaking up sitting time reduces cardiometabolic risk markers. The aim of this study is to therefore observe if this effect is replicated in the cardiac population and thus whether breaking up sitting time will reduce the risk of a secondary cardiac event.

Potential participants will be required to meet an inclusion criteria to take part in the study: aged 50 years or above and had a myocardial infarction within the past three months at the time of recruitment to the study.

Participants will be randomised to each condition: 1) uninterrupted sitting; 2) sitting with intermittent standing and 3) sitting with intermittent light physical activity (stepping to a metronome beat). A number of physiological markers will be measured before, during and after each condition and analysed to compare the effectiveness of each condition.

All measurements will be taken at the University of Bedfordshire Sport and Exercise Science Laboratories.

DETAILED DESCRIPTION:
Study design A repeated measures, randomised cross over study design will be used. All data collection will take place at the Sport and Exercise Science Laboratories, University of Bedfordshire, Polhill Avenue, Bedford, UK. After a preliminary testing session, participants will complete three, 6-hour experimental conditions in a random order: 1) uninterrupted sitting; 2) sitting interrupted with standing breaks, and 3) sitting interrupted with light intensity stepping breaks. There will be a washout period of at least 72 hours between conditions, as previous research suggests that a single session of exercise can affect blood glucose levels for the following 48 hours (Mikines, et al., 1988). Participants will be randomised to order of condition using computer generated random numbers. This will assign them a trial order using block randomization with balanced block sizes. Participants will be blinded to the trial condition until they arrive on the day of their first and second experimental conditions.

Preliminary testing Patients will first attend a preliminary testing session where they will become accustomed to light intensity stepping on the spot to the beat of a metronome and use of the Borg RPE scale. This will ensure patients are familiar with an intensity that is equivalent to an RPE of 8-11 (very light to light) that will be used in the respective experimental condition. Participants will step to different metronome paces starting at a slow pace and building up gradually every 1-2 minutes until an RPE of 8-11 is found. This imitates the intensity recommended within the warm up of CR, as recommended by BACPR. Height (cm) and weight (kg) will also be measured using a stadiometer (Harpenden 98.602, Holtain Ltd., Crymych) and digital scales (Tanita BWB0800, Tanita Corp., Tokyo, Japan) respectively, to calculate body mass index (kg/m2).

Experimental Protocol Participants will be asked to refrain from any alcohol and caffeine for 24 hours prior to each visit, as well as avoid exercise for 72 hours and complete an overnight fast. This will be explained to them during the preliminary visit. To monitor this, they will be asked prior to participation per visit whether they have fasted/ when they last ate and drank.

Participants will be asked to perform an overnight fast for at least 10 hours before arrival and minimise active travel to the laboratory (e.g. use a car for travel). They will rest for 30 minutes to achieve a steady state before baseline blood pressure (two measures with 2 minutes rest between each and the average taken) and blood samples are taken. Baseline cardiac function measures (global strain, ejection fraction and systolic volume) will be measured using an echocardiogram scan, as well as an electrocardiogram (ECG) to ensure there are no electrical contraindications to the heart which would make the participant unsuitable to complete the study intervention including ST depression / elevation or any arrythmias. Baseline mood and wellbeing measures will then be assessed using questionnaires.

Following baseline measures, a standardised breakfast will be consumed (see meals section below) and participants will then commence the experimental condition. See Figure 1 for schematic of experimental conditions.

The three experimental conditions for this study are:

1. Uninterrupted sitting for 6 hours.
2. Sitting interrupted with 5 minutes of static standing every 30 minutes.
3. Sitting interrupted with 5 minutes of light intensity stepping every 30 minutes using a metronome at the intensity determined during preliminary testing. This replicates active recovery time currently performed in a phase III CR class.

A lunch meal will be provided at 12:00 during each condition. During sitting periods, participants will be able to read books, magazines or newspapers and/or watch TV, DVDs or media streaming services. Participants will be transported to the toilets and food consumption areas using a wheelchair to ensure activity is minimised and standardised between conditions.

Standardised food and water intake Each meal will provide approximately 30% of estimated daily energy requirements. This will be calculated for each individual participant using a prediction equation based on individual's height, weight and gender. Breakfast will consist of bran flakes, whole milk, and a honey and granola bar and will consist of 54% carbohydrate, 34% fat and 12% protein. Lunch will consist of a chicken sandwich, salted crisps and jammie dodger biscuit (54% carbohydrate, 34% fat and 12% protein). The macronutrient composition of the meals are in general agreement with guidelines recommended for a balanced diet (Public Health England, 2016). Participants will be encouraged to consume their meal within 15 minutes. The time taken will be recorded in the first condition and this time will then be replicated in the latter two conditions. Water will be available for the participants ad libitum during their first experimental condition visit. This volume of intake will be recorded and the same amount provided in the following two conditions spread over the day.

Data collection Finger prick capillary whole blood samples will be collected at baseline, 30, 60, 120, 180, 210, 240, 300 and 360 minutes throughout the conditions to allow later analysis of glucose, triglycerides, HDL-C, and insulin. Blood samples will be taken after the hand is pre-warmed in warm water for approximately 5 minutes. Blood pressure and heart rate will be measured 5 minutes before each of the blood samples are taken. Cardiac function measures and mood and wellbeing will be measured at baseline and post-condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients post myocardial infarction (ST wave elevated MI or Non-ST wave elevated MI) within the past three months (confirmed by elevated blood biomarkers or electrocardiographic changes), in which the procedure/ recovery uncomplicated and are therefore classified as low risk.
* Aged 40 years or above.
* Any ethnicity.
* Individuals with diet controlled type 2 diabetes mellitus

Exclusion Criteria:

* Previous MI
* Under 40 years of age.
* Unable to provide valid informed consent (lack of mental capacity).
* Not had a cardiac event diagnosed within the past three months.
* Existing comorbidities including cancer, chronic kidney disease and gastro-oesophageal diseases.
* Unstable coronary disease.
* Diagnosed diabetes and use of medication.
* Disease or conditions with a prognosis of less than 6 months to end of life (palliative care). Any known blood borne disease.
* Unable to stand and engage in light-intensity stepping.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Posterior wall thickness | 4 months
  Posterior wall thickness in cm
Interventricular septum | 4 months
  Interventricular septum in cm
Left ventricular internal diameter | 4 months
  Left ventricular internal diameter in cm
Aortic root | 4 months
  Aortic root in cm
End volume | 4 months
  End volume in cm
E wave | 4 months
  E wave in ms
A wave | 4 months
  A wave in ms
Relative wall thickness | 4 months
  Relative wall thickness in cm
Left ventricular mass | 4 months
  Left ventricular mass in g
E/A ratio | 4 months
  E/A ratio
Deceleration time | 4 months
  Deceleration time in ms
Isovolumetric relaxation time | 4 months
  Isovolumetric relaxation time in ms
Ejection fraction | 4 months
  Ejection fraction in %
Stroke volume | 4 months
  Stroke volume in L

SECONDARY OUTCOMES:
Systolic Blood pressure | 4 months
  Resting systolic blood pressure in mmHg
Diastolic Blood pressure | 4 months
  Resting diastolic blood pressure in mmHg
Postprandial triglycerides | 4 months
  Postprandial triglycerides in mmol/L
Postprandial total cholesterol | 4 months
  Postprandial total cholesterol in mmol/L
Postprandial low density lipoprotein cholesterol | 4 months
  Postprandial low density lipoprotein cholesterol in mmol/L
Postprandial high density lipoprotein cholesterol | 4 months
  Postprandial high density lipoprotein cholesterol in mmol/L
Postprandial insulin | 4 months
  Postprandial insulin in mU/L
Postprandial glucose | 4 months
  Postprandial glucose in mmol/L
Mood and wellbeing | 4 months
  Positive affect and negative affect scale. This is a 5 point score, that asks 10 questions about positive feelings and 10 questions about negative feelings. The higher the score for each scale, the more likely they are feeling positive or negative.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Richards, PhD, Study Director — University of Bedfordshire; Abbie C Bell, MSc, Principal Investigator — Bedfordshire Hospitals NHS Foundation Trust
Locations (1):
- Cardiac Rehabilitation, Bedford, Bedfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Upon registration to the study, participants will be given a unique participant ID number, which will henceforth be used in all data collection within the study. This will be determined using a number system. A confidential log will be kept by the research team to identify participants with their anonymous ID numbers, which will be encrypted on a secure computer. All other electronic documentation will also be encrypted. Only direct members of the research team will have access to the data, and will be listed on the study's delegation log. Where data is transmitted to sponsors, if necessary, it will only be identifiable by its participant ID number, thus not becoming patient identifiable at any time.

DOCUMENTS (1):
  • Study Protocol (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/75/NCT05193175/Prot_000.pdf